CLINICAL TRIAL: NCT00485667
Title: Evaluation of the Effects of Therapeutic and Supra-therapeutic Single Doses of SKY0402 Given as Subcutaneous Injection on the QT/QTc Interval in Young Healthy Volunteers. A Prospective, Randomized, Placebo- and Positive-controlled, Double Blind, Single-centre, Crossover Phase 1 Study.
Brief Title: Phase 1 Thorough QT Study in Young Healthy Volunteers
Acronym: TQT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Collaborators: Richmond Pharmacology Limited (Industry)
Responsible Party: Dr. Jorg Taubel, Richmond Pharmacology Ltd
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SKY0402C105; Richmond No. C07027; EudraCT Number: 2007-001981-33
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Postoperative Pain
Keywords: pain; postoperative
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Moxifloxacin tablet (Active Comparator)
  Interventions: Drug: SKY0402; Drug: Moxifloxacin 400mg; Drug: Placebo injection
- Placebo tablet (Experimental)
  Interventions: Drug: SKY0402; Drug: Placebo injection; Drug: Placebo tablet
- SKY0402 300mg (Experimental)
  Interventions: Drug: SKY0402; Drug: Moxifloxacin 400mg; Drug: Placebo tablet
- SKY0402 450mg (Experimental)
  Interventions: Drug: SKY0402; Drug: Moxifloxacin 400mg; Drug: Placebo tablet
- Placebo injection (Placebo Comparator)
  Interventions: Drug: Moxifloxacin 400mg; Drug: Placebo injection; Drug: Placebo tablet

INTERVENTIONS:
Drug: SKY0402 — Subects received either 300mg or 450mg
  Arms: Moxifloxacin tablet; Placebo tablet; SKY0402 300mg; SKY0402 450mg
Drug: Moxifloxacin 400mg
  Arms: Moxifloxacin tablet; Placebo injection; SKY0402 300mg; SKY0402 450mg
Drug: Placebo injection
  Arms: Moxifloxacin tablet; Placebo injection; Placebo tablet
Drug: Placebo tablet
  Arms: Placebo injection; Placebo tablet; SKY0402 300mg; SKY0402 450mg

SUMMARY:
A reduction in the postoperative need for opioids to enhance the recovery process and increase patient postoperative satisfaction.

DETAILED DESCRIPTION:
Providing extended pain relief without the use of indwelling catheters is the basis for developing SKY0402. A formulation of bupivacaine, given as a single injection after surgery, that could provide adequate, continuous, and extended pain relief would greatly simplify postoperative pain management, reduce the need for repeated administration, and minimize break-through episodes of pain.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult Caucasian men or non-pregnant, non-lactating women between 18 and 40 years of age, inclusive.
2. Healthy as judged by responsible physician with no clinically significant abnormality identified on the medical and laboratory evaluation, including 12-lead ECG and vital signs.
3. Non-smoker in the previous 3 months.
4. Body weight greater than or equal to 50 kg and BMI within the range 19-29 kg/m2, inclusive.
5. At screening and Run-in period each ECG should have:

   * Consistent sinus rhythm, (i.e. if greater than or equal to 2 ECGs are not sinusal at different time points the volunteer should not be included),
   * No clinically significant conduction disorder,
   * PR between 120 and 230 ms,
   * HR less than or equal to 100 beats/min and greater than or equal to 40 beats/min,
   * QRS < 120 ms,
   * QT intervals that can be consistently analysed,
   * QTcB less than or equal to 430 ms for males,
   * QTcB less than or equal to 450 ms for females

   If there are outlying values in the ECGs, the consistency of these values should be confirmed as follows:
   * If HR is between 40 and 44 bpm (inclusive) in 2 ECGs (of one triplicate) on more than one time point during Run-in, subject should not be selected. Conversely, this means that if HR is between 40 and 44 bpm at screening and/or on just one time-point-triplicate during Run-in, the volunteer can be selected.
   * If HR < 40 bpm on a single occasion at screening or in Run-in period, subject should not be selected,
   * If PR interval is consistently out-of-range (< 120 or > 230 ms) during Run-in period, i.e. in 2 out of 3 ECGs at one time point or in one ECG at more than one time point, the cardiologist needs to perform a manual measurement of this value. If the manual measurement confirms that PR is out-of-range, the volunteer must not be selected.
   * If QRS is consistently >120 ms during run-in period, i.e. in 2 ECGs of a triplicate or in 2 ECGs from 2 different time-points, the cardiologist needs to perform a manual measurement of this value. If the manual measurement confirms the QRS is out-of-range, the volunteer must not be selected.
   * If QTcB is out of range (QTcB >430 ms for males or >450 ms for females, or repeated demonstration of a QTcB interval >440 ms for females) even on a single occasion, it should be checked whether the heart rate is constant. If the HR is not constant and if the increase in QTcB is clearly due to hysteresis (e.g. on the immediate repeated ECG with consistent HR the QTcB is back to normal), then the volunteer can be selected. If the HR is constant and the QTcB is still out-of-range, the cardiologist needs to perform a manual measurement and calculation of the QTcB. If the QTcB is normal on manual measurement, the volunteer can be selected. If the QTcB is abnormal on manual measurement without acceptable cause, the volunteer must not be selected, even if the QTcB is outlying on one single ECG.

   The final decision to include / not include a volunteer based on protocol ECG criteria lies with the cardiologist assessing the Run-in ECGs.
6. Signed and dated written informed consent prior to admission to the study.
7. The subject is able to understand and comply with protocol requirements, instructions, and protocol-stated restrictions.
8. A female subject may be entered into the study if she is:

   * Post-menopausal female defined as being amenorrhoeic for greater than 2 years with an appropriate clinical profile, e.g. appropriate age and history of vasomotor symptoms. However; if indicated, this should be confirmed by estradiol and FSH levels consistent with menopause (according to local laboratory ranges).
   * Pre-menopausal females with a documented hysterectomy (medical report verification) and/or bilateral oophorectomy. In the case of oophorectomy alone, only acceptable when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
   * Females of childbearing potential must use one of the following methods of contraception:

     * Abstinence
     * Surgical sterilisation (tubal ligation)
     * use oral contraceptives, injectable progesterone, or subdermal implants
     * use double barrier method consisting of spermicide in addition to using a condom, or having another form of contraception such as an intrauterine device, diaphragm, or cervical cap.

Exclusion Criteria:

1. History or presence of clinically significant haematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease.
2. History of clinically significant syncope.
3. Family history of sudden death.
4. Family history of premature cardiovascular death.
5. Clinically significant history or family history of congenital long QT syndrome (e.g. Romano-Ward syndrome, Jervell and Lange-Nielson syndrome) or Brugada's syndrome.
6. History of clinically significant arrhythmias (especially ventricular arrhythmias, atrial fibrillation, or recent conversion from atrial fibrillation).
7. Complete bundle branch block / sinus node dysfunction.
8. Conditions predisposing the volunteer to electrolyte imbalances (e.g. altered nutritional states, chronic vomiting, anorexia nervosa, bulimia nervosa).
9. Any pathology or abnormality with possible influence on the ECGs.
10. Clinically significant dermatological disease including history of drug-induced skin rash.
11. History of clinically significant psychiatric illness.
12. History of gastro-intestinal surgery except appendectomy, herniotomy and cholecystectomy.
13. History of chronic inflammation of gastro-intestinal tract.
14. History of tendinopathy with fluoroquinolone.
15. Subjects with vital signs measurements as follows:

    * Supine heart rate outside the 40 to 100 beats/min range,
    * Standing heart rate outside the 40 to 125 beats/min range,
    * Supine systolic blood pressure outside the 80 to 140 mmHg range
    * Supine diastolic blood pressure outside the 40 to 95 mmHg range.
16. Subjects with a symptomatic drop in systolic blood pressure of > 20 mmHg and diastolic > 10 mmHg at screening.
17. A positive pre-study HIV 1 & 2 antibodies, Hepatitis B surface antigen, and/or Hepatitis C antibody result.
18. Positive serum pregnancy tests for women of childbearing potential.
19. Subjects with a confirmed positive pre-study urine drugs of abuse / alcohol breath test.
20. History or evidence of drug or alcohol abuse within 18 months of study start.
21. Abuse of alcohol defined for males as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units; or for females defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units. One unit is equivalent to a half-pint(220 mL) of beer or 1 (25 ml) measure of spirits or 1 glass (125 ml) of wine.
22. Use of prescribed medication during the two weeks before the baseline ECG day in Period 1 and use of OTC drugs (including herbal remedies and minerals) in the week before the baseline ECG day in Period 1 (or 14 days if the drug has enzyme affecting properties), unless in the opinion of the Investigator and Sponsor the medication will not interfere with the study procedures or compromise subject safety. Use of medications which are known to carry a risk of causing Torsades de Pointes is not allowed within 14 days or 10 times the elimination half life (whichever is longer) before the baseline ECG day in Period 1. Use of vitamins is not allowed within 48 hours before the baseline ECG day in Period 1. Oral contraceptive drugs for women of childbearing potential and occasional use of paracetamol (up to 2 g/day) for pain and fever relief is allowed.
23. History or presence of allergy to the study drugs or drugs in their respective classes, or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation.
24. A known history of hypersensitivity to drugs, specifically to any component of the study medication, or history of hypersensitivity to moxifloxacin or any member of the quinolone class of antimicrobial agents.
25. The subject has eaten grapefruit, grapefruit juice, Seville oranges, watercress, broccoli, brussel sprouts or cabbage within seven days before the baseline ECG day in Period 1.
26. Participation in a study with an investigational drug within 90 days prior to the baseline ECG day in Period 1.
27. Blood donation or blood loss within 90 days prior to the baseline ECG day in Period 1.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2007-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
ECG findings using the best heart rate correction method | Up to 96 hours

SECONDARY OUTCOMES:
QT/QTc interval data variations from baseline | up to 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jorg Taubel, MD MFPM, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology Ltd, London, United Kingdom